CLINICAL TRIAL: NCT05673330
Title: Effects of Spinal Mobilization Versus Myofacial Release Techniques on Pain And Disability In Patients With Tension Type Headache
Brief Title: Spinal Mobilization Versus Myofacial Release Techniques On Pain And Disability In Patients With Tension Type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AH/22/Faryall Kemall
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Tension Type Headache
Keywords: Tension Type Headache
MeSH Terms: conditions — Tension-Type Headache | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Mobilizations (Active Comparator): 1. Headache SNAG: A posteroanterior mobilization of the second cervical vertebrae is sustained for 10 to 30 s with the aim to reduce headache intensity at the time of application. (6)
  2. Maitland's C1-C7 PA Glide: A posteroanterior (PA) mobilization of the first till seventh cervical vertebra is achieved by applying a force on to a vertebral segment in a posteroanterior direction (Back to front).
  The patients will receive Spinal Mobilizations consisting of 1 set of 6 repetitions once daily thrice per week for four weeks. Pre and post intervention values will be taken on 1st day and after 4 weeks.
  Interventions: Other: Spinal Mobilizations
- Myofascial Release technique (Active Comparator): Suboccipital Inhibition Technique: While the patient will be in the supine position, the physician sitting at the top end of the table will place the fingers of both hands on the patient's suboccipital region. Flexi-perpendicular long fingers exerting an inhibitory pressure on the muscle insertions of the neck extensors in the occiput, perpendicularly to muscle fibers, while the thumbs counterbalance the head against rotation. A deep and progressive pressure would be applied perpendicular to the fibers until a decrease in muscle tone would be detected. This deep and progressive pressure would be maintained for a total of 10 min until release of suboccipital tissues is achieved.
  The patients will receive myofascial release with the frequency of 1 set and 10 repetitions once a day three times per week for four weeks. Pre and post intervention values will be taken on 1st day and after 4 weeks.
  Interventions: Other: Myofascial Release Technique

INTERVENTIONS:
Other: Spinal Mobilizations — 1. Headache SNAG: A posteroanterior mobilization of the second cervical vertebrae is sustained for 10 to 30 s with the aim to reduce headache intensity at the time of application. (6)
  2. Maitland's C1-C7 PA Glide: A posteroanterior (PA) mobilization of the first till seventh cervical vertebra is achieved by applying a force on to a vertebral segment in a posteroanterior direction (Back to front).
  The patients will receive Spinal Mobilizations consisting of 1 set of 6 repetitions once daily thrice per week for four weeks. Pre and post intervention values will be taken on 1st day and after 4 weeks
  Other Names: Headache SNAG, Maitland's C1-C7 PA Glide
  Arms: Spinal Mobilizations
Other: Myofascial Release Technique — Suboccipital Inhibition Technique: While the patient will be in the supine position, the physician sitting at the top end of the table will place the fingers of both hands on the patient's suboccipital region. Flexi-perpendicular long fingers exerting an inhibitory pressure on the muscle insertions of the neck extensors in the occiput, perpendicularly to muscle fibers, while the thumbs counterbalance the head against rotation. A deep and progressive pressure would be applied perpendicular to the fibers until a decrease in muscle tone would be detected. This deep and progressive pressure would be maintained for a total of 10 min until release of suboccipital tissues is achieved.
  The patients will receive myofascial release with the frequency of 1 set and 10 repetitions once a day three times per week for four weeks. Pre and post intervention values will be taken on 1st day and after 4 weeks.
  Other Names: Suboccipital Inhibition Technique
  Arms: Myofascial Release technique

SUMMARY:
The most frequent kind of primary headache is tension headache, often known as stress headache or tension-type headache (TTH). The pain usually affects both sides of the head and might extend from the lower back of the head, the neck, the eyes, or other muscle groups in the body. Nearly 90 percent of all headaches are tension-type headaches causing a debilitating effect on job productibility and overall quality of life. The aim of the study will be to compare the effects of spinal mobilizations comprising Mulligan's headache SNAGs and Maitland's PA glide with the myofascial release technique on pain and disability in patients with tension-type headache.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at FMH Physiotherapy Clinic, NUR International Physical Therapy clinic and Boston Physiotherapy Clinic Lahore through consecutive sampling technique on 34 patients which will be allocated using simple random sampling through sealed opaque envelopes into Group A and Group B. Group A will be treated with Spinal Mobilizations comprising Mulligan's headache SNAGs and Maitland's PA glide and Group B will be treated with Myofascial release technique. Outcome measures tools will be conducted through NPRS, Headache disability Index, Headache impact test (HIT-6). Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups

ELIGIBILITY:
Inclusion Criteria:

* • Male and female between ages of 30-60 years

  * Presence of 2 or more of the following: bilateral headache, pressure or squeezing pain, mild or intermediate pain intensity, and headache not elicited by daily physical activities
  * Headache lasting between 30 minutes and 7 days
  * Patients with no increase in pain during physical activity
  * Patients not having any photophobia, phonophobia during headache
  * Headache unaccompanied by vomiting or nausea

Exclusion Criteria:

* Any other primary or secondary headache according to the ICHD-III criteria.

  * A history of neck or head trauma (e.g., whiplash).
  * Any red flags (vertebral tumor, fracture, dislocation and infection, metabolic diseases, rheumatic and connective tissue diseases, systemic neuromuscular diseases, prolonged history of steroid use).
  * Diagnosis of any structural spinal disorders (osteoporosis, disc herniation, myelopathy, spinal stenosis, spondylolisthesis).
  * Prior surgery to the cervical spine.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
International Classification of Headache Disorders Criteria (ICHD-3 beta) | 4 weeks
  It is used for diagnosis of the tension type headache and has following specifications: The pain should be bilateral, pressing and tightening pain, having a mild-moderate intensity [≤7.0 on a visual analog scale (VAS)] and there should be no increase in pain with physical activity. The patients should not have phonophobia, nausea, vomiting or photophobia. Headache should last between 30 minutes and 7 days
Numeric pain rate scale (NPRS) | 4 weeks
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain"
Headache Disability Index Questionnaire | 4 weeks
  To quantify the impact of headache on daily living, a 25-item headache disability inventory (HDI) will be used. Each requiring a "yes" (four points), "sometimes" (two points), or "no" (zero points) response based on items derived empirically from case history responses of subjects with headache. Items are sub grouped into functional and emotional subscales
Headache Impact Test (HIT-6) | 4 weeks
  The HIT-6 is a 6-item screening instrument used to quantify headache. It assesses the effects of headaches on daily life activities. This questionnaire has 6 questions, with a maximum number of points of 6*13 (78). A total score of 36 means best and 78 means worst in terms of headache. Scores above 50 are "high".

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Study Principal Investigator
Locations (1):
- NUR International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corum M, Aydin T, Medin Ceylan C, Kesiktas FN. The comparative effects of spinal manipulation, myofascial release and exercise in tension-type headache patients with neck pain: A randomized controlled trial. Complement Ther Clin Pract. 2021 May;43:101319. doi: 10.1016/j.ctcp.2021.101319. Epub 2021 Jan 24. PMID 33517104
- [Background] Zhang Y, Kong Q, Chen J, Li L, Wang D, Zhou J. International Classification of Headache Disorders 3rd edition beta-based field testing of vestibular migraine in China: Demographic, clinical characteristics, audiometric findings and diagnosis statues. Cephalalgia. 2016 Mar;36(3):240-8. doi: 10.1177/0333102415587704. Epub 2015 May 18. PMID 25986149
- [Background] Akbas I, Kocak AO, Akgol Gur ST, Oral Ahiskalioglu E, Dogruyol S, Dolanbay T, Demir M, Cakir Z. Lidocaine versus dexketoprofen in treatment of tension-type headache: A double-blind randomized controlled trial. Am J Emerg Med. 2021 Mar;41:125-129. doi: 10.1016/j.ajem.2020.12.057. Epub 2021 Jan 7. No abstract available. PMID 33423013
- [Background] GBD 2016 Headache Collaborators. Global, regional, and national burden of migraine and tension-type headache, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):954-976. doi: 10.1016/S1474-4422(18)30322-3. PMID 30353868
- [Background] Schiller J, Karst M, Kellner T, Zheng W, Niederer D, Vogt L, Eckhardt I, Beissner F, Korallus C, Sturm C, Egen C, Gutenbrunner C, Fink MG. Combination of acupuncture and medical training therapy on tension type headache: Results of a randomised controlled pilot study. Cephalalgia. 2021 Jul;41(8):879-893. doi: 10.1177/0333102421989620. Epub 2021 Feb 9. PMID 33563049
- [Background] Satpute K, Bedekar N, Hall T. Effectiveness of Mulligan manual therapy over exercise on headache frequency, intensity and disability for patients with migraine, tension-type headache and cervicogenic headache - a protocol of a pragmatic randomized controlled trial. BMC Musculoskelet Disord. 2021 Mar 3;22(1):243. doi: 10.1186/s12891-021-04105-y. PMID 33657998
- [Background] Pourahmadi M, Dommerholt J, Fernandez-de-Las-Penas C, Koes BW, Mohseni-Bandpei MA, Mansournia MA, Delavari S, Keshtkar A, Bahramian M. Dry Needling for the Treatment of Tension-Type, Cervicogenic, or Migraine Headaches: A Systematic Review and Meta-Analysis. Phys Ther. 2021 May 4;101(5):pzab068. doi: 10.1093/ptj/pzab068. PMID 33609358
- [Background] Osama M. Effects of autogenic and reciprocal inhibition muscle energy techniques on isometric muscle strength in neck pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2021;34(4):555-564. doi: 10.3233/BMR-200002. PMID 33523036
- [Background] Kwon SH, Chung EJ, Lee J, Kim SW, Lee BH. The Effect of Hamstring Relaxation Program on Headache, Pressure Pain Threshold, and Range of Motion in Patients with Tension Headache: A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Sep 27;18(19):10137. doi: 10.3390/ijerph181910137. PMID 34639438
- [Background] Choi W. Effect of 4 Weeks of Cervical Deep Muscle Flexion Exercise on Headache and Sleep Disorder in Patients with Tension Headache and Forward Head Posture. Int J Environ Res Public Health. 2021 Mar 25;18(7):3410. doi: 10.3390/ijerph18073410. PMID 33806089